**Title: Pilot Study:** Clinical assessment of bipolar radiofrequency microneedling for improved and wrinkled of the suprapatellar skin.

NCT Number: NCT03507036

IRB Approval Date: 28 AUGUST 2018

## Statistical Analysis Plan

Statistical analysis was performed using GraphPad Prism (Version 7, GraphPad Inc.; San Diego, CA, USA). One-sample t-tests were used to evaluate the percent change from baseline (before treatment or untreated skin) of the non-invasive skin assessments at both 3 weeks and 6 months post ablation. Statistical significance was determined by a p < 0.05.